CLINICAL TRIAL: NCT05512455
Title: Comparison of the Precision of the Virtual Articulators Using Various Virtual Articulator Mounting Procedures
Brief Title: Accuracy of Various Virtual Articulator Mounting Procedures: An in Vivo Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Hao Yu, Fujian Medical University, Fujian Medical University
Other Study IDs: 2022071901
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Occlusion
Keywords: virtual articulator ,occlusion
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- virtual articulator mounting using an average facebow: indirect virtual mounting in MS VA by using an average facebow
- virtual articulator mounting by using average values: virtual mounting in MS VA by using average values;
- virtual articulator mounting by using professional facial scanner: virtual mounting in MS VA by using professional facial scanner
- virtual articulator mounting by using smartphone facial scanner: virtual mounting in MS VA by using smartphone facial scanner
- virtual articulator mounting by using CBCT located in Bergstrom's point: virtual mounting in MS VA by using CBCT located in Bergstrom's point
- virtual articulator mounting by using CBCT located in the medial poles of the condyle: virtual mounting in MS VA by using CBCT located in the medial poles of the condyle
- virtual articulator mounting by using JMA: virtual mounting in CA VA by using JMA,as the group to compare with the other mounting procedures.

SUMMARY:
the aim of this study was to evaluate the accuracy of the various virtual articulator mounting procedures.

DETAILED DESCRIPTION:
The purpose of the present study was to evaluate the accuracy of various virtual articulator mounting procedures. For this purpose, 7 kinds of virtual mounting procedures were investigated:(1) indirect virtual mounting in MS VA by using an average facebow; (2) virtual mounting in MS VA by using average values; (3) virtual mounting in MS VA by using professional facial scanner; (4) virtual mounting in MS VA by using smartphone facial scanner; (5) virtual mounting in MS VA by using CBCT located in Bergstrom's point; (6) virtual mounting in MS VA by using CBCT located in the medial poles of the condyles; (7) virtual mounting in CA VA by using JMA，as the group to compare with the other mounting procedures. The null hypothesis is that no difference would be found in the static measurements taken virtually when comparing these 7 procedures for virtual mounting.

ELIGIBILITY:
Inclusion Criteria:

* 1.without any symptoms and signs of the temporomandibular joint 2.Willing to participate and to sign a written informed consent form 3.in good health and had no past history of any serious illness

Exclusion Criteria:

* emporomandibular or craniocervical disorders

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: 10 females and 10 males
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-20 (Estimated)

PRIMARY OUTCOMES:
the accuracy of different virtual articulator mounting procedures | immediately
  the virtual articulator mounting by using JMA is considered as the the gold standard, which can calculate the hinge axis of the temporomandibular joint, compare the hinge axis of the temporomandibular joint of different virtual articulator mounting procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Yu, Principal Investigator — Fujian Medical University
Locations (1):
- Fujian Medical University, Fuzhou, Fujian, China